CLINICAL TRIAL: NCT00458016
Title: A Phase 2, 28-day, Multicenter, Double-Blind,Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability and Efficacy of MB07803 in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerability, and Efficacy Study of MB07803 Administered to Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB07803-202
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: MB07803
- 2 (Experimental)
  Interventions: Drug: MB07803
- 3 (Experimental)
  Interventions: Drug: MB07803
- 4 (Experimental)
  Interventions: Drug: MB07803
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MB07803 — Daily oral administration
  Arms: 1; 2; 3; 4
Drug: Placebo — Daily oral administration
  Arms: 5

SUMMARY:
The purpose of this study is to collect important information regarding the safety, tolerability, and efficacy of MB07803 when administered for 28 days in patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose between 120 - 270 mg/dL at screening
* HbA1c measurements between 6.0 - 10% at screening
* Females who are surgically sterile (i.e. women who have had a hysterectomy or tubal ligation). Females who are postmenopausal for at least 12 consecutive months and documented by blood follicular stimulating hormone (FSH) greater than or equal to 40 mlU/mL.Females of childbearing potential must be willing to use an approved double-barrier method of birth control (e.g. condom plus spermicide ;IUD plus spermicide) from the time of signing the informed consent form through 4 weeks following the last dose of study drug.
* Body mass index (BMI) in the range of 18.5 - 37 kg/m2 Patients with a BMI in the range of 37.5 - 40 kg/m2 who in the Investigator's opinion, are in good health and satisfy the eligibility criteria, will be considered on a case-by case basis
* Written informed consent

Exclusion Criteria:

* Type 1 diabetes mellitus
* Type 2 diabetes mellitus with a history of diabetic ketoacidosis or ketosis-prone
* Use of thiazolidinediones (TZDs)
* Currently on more than two oral hypoglycemic agent
* History of outpatient insulin use
* Clinically significant history of cardiac disease within 6 months of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma Glucose Concentration | Change from baseline to Day 28

SECONDARY OUTCOMES:
Fasting serum triglycerides and free fatty acids, fasting serum insulin. | Change from baseline to Day 28

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Los Angeles, California
  - Walnut Creek, California
  - Miami, Florida
  - Miami Gardens, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Butte, Montana
  - Las Vegas, Nevada
  - Charlotte, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Delaware, Ohio
  - Marion, Ohio
  - Willoughby Hills, Ohio
  - Tulsa, Oklahoma
  - Charleston, South Carolina
  - Bristol, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia